CLINICAL TRIAL: NCT06798142
Title: Risk Stratification and Heterogeneity for Organ Damage in Acute Diquat Poisoning: A Multi-Center Cohort Study
Brief Title: Risk Stratification and Heterogeneity for Organ Damage in Acute Diquat Poisoning
Status: Active, not recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hao Sun, Principal Investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: 2025-1047-02
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Toxic Encephalopathy; Diquat Poisoning
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — plasma

INTERVENTIONS:
Procedure: extracorporeal treatment — Extracorporeal treatments included hemoperfusion (HP) and continuous veno-venous hemodiafiltration (CVVHDF).

SUMMARY:
This study aims to characterize the relationship between plasma diquat concentrations and organ damage risk.

ELIGIBILITY:
Inclusion criteria:

1. history of oral exposure to diquat solution reported by patient or proxy;
2. a specimen for the diquat plasma concentration collected immediately upon admission;
3. documentation that patients or, in case of unconsciousness of the patient, legal proxies were aware of and agreed to treatment plans.

Exclusion criteria:

1. they had ingested other toxins in addition to diquat (qualitative toxicological screening tests);
2. diquat was not detected in specimens, or plasma concentration data were unavailable;
3. patients with an exposure time (time from exposure to emergency department presentation) longer than 48 hours;
4. data on organ damage were not unavailable;
5. combined with other central nervous system injuries other than toxic encephalopathy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with the history of acute diquat poisoning
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival outcome | 28 days within the index date of presentation at emergency department

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China